CLINICAL TRIAL: NCT02335463
Title: 3D Single Cell Analysis Using Cell Morphology and Organelle Scattering Texture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201402039RINB
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Cancer
Keywords: optical coherence tomography
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will use an advanced high resolution 3D optical coherence tomography (OCT) technology to observe colon and skin images in ex vivo.

DETAILED DESCRIPTION:
Achieved formalin-fixed paraffin embedded tissue specimens from colon cancers and/or other benign and pre-cancer colon lesions as well as melanoma and/or other benign pigmented skin lesions will be used. The achieved specimens were kept in Department of Pathology, National Taiwan University Hospital. Sections of achieved pathological specimens were put on glass slides and tissue image will be observed by 3D optical coherence tomography (OCT). The 3D optic tomography system utilize a Ce:YAG optical fiber as light source and also combined with confocal microscopy. Taken together, these features made the 3D optic tomography system have very high resolution and suitable for single cell imaging. This study will not interfere with the normal medical practice and had no impact on patient's safety and health. All of the materials will be destroyed once the experiments are done. The enrollment criteria will be patients who underwent colon/skin surgery or examinations in NTUH with pathological specimens taken and stored at NTUH.

ELIGIBILITY:
Inclusion Criteria:

• Participants are those who who received skin or colon surgery, with their surgical specimens preserved and stored at Department of Pathology, National Taiwan University Hospital.

Exclusion Criteria:

• Age younger than 20 years old.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are those who received skin or colon surgery, with their surgical specimens preserved and stored at Department of Pathology, National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Image of colon or skin tissue | 1 day
  Image of colon or skin tissue

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Lung HUANG, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan